CLINICAL TRIAL: NCT00002994
Title: A Pilot Study of Low-Dose Interleukin-2 Plus Recombinant Human Anti-HER2 Monoclonal Antibody in Solid Tumors
Brief Title: Interleukin-2 Plus Monoclonal Antibody Therapy in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9661; CLB-9661; CDR0000065541 (Registry Identifier: NCI Physician Reference Desk)
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Monoclonal antibody + interleukin 2 (Experimental): Cycle 1: low dose IL2 days 1-7; MoAb day 7; intermediate dose IL-2 days 8-10; Low dose IL2 days 11-20.
  Cycle 2 & all subsequent cycles: MoAb day 1; intermediate dose IL2 days 1-3; low dose IL2 days 4-14
  Interventions: Biological: interleukin 2; Biological: rhuMAb

INTERVENTIONS:
Biological: interleukin 2 — low dose: 1 million IU/square meter subq injection q day days 1-7 and 11-20 cycle 1; days 4-14 subsequent cycles Intermediate dose: 12 million IU/square meter subq injection on days 8-10 of cycle 1; days 1-3 of subsequent cycles
Biological: rhuMAb — 90 min IV infusion day 7 of each cycle

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill solid tumor cells. Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Pilot study to examine the effectiveness of interleukin-2 plus monoclonal antibody in treating patients who have solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxic effects of humanized anti-HER2 monoclonal antibodies when administered in combination with interleukin-2 (IL-2) in patients with solid tumors. II. Measure in vitro cytotoxicity using peripheral blood mononuclear cells, plasma, and target cell lines that express HER2 in this patient population. III. Phenotypically characterize effector cells at the time of antibody administration and 24 hours after three days of intermediate dose IL-2 pulsing in these patients. IV. Measure antitumor response in these patients.

OUTLINE: Cohorts of 6 patients are enrolled at 4 antibody dose levels. After at least 6 patients have been treated on study for at least 30 days, the next dose level may be initiated provided that fewer than 2 of the first 6 evaluable patients experience dose limiting toxicity (DLT) related to either the antibody or the combination of antibody with interleukin-2 (IL-2). If 2 or more patients experience DLT, the next cohort is enrolled at the antibody dose midway between the current and previous dose levels. An additional 6 patients are entered at the maximum tolerated dose. On course 1, patients receive IL-2 subcutaneously (SQ) daily on days 1-7 and humanized anti-HER-2 monoclonal antibodies IV over 90 minutes on day 7. Patients receive intermediate dose pulsed IL-2 SQ on days 8-10 and low dose IL-2 SQ on days 11-20. On course 2 and all subsequent courses, patients receive humanized anti-HER2 monoclonal antibodies IV immediately prior to IL-2 (SQ) on day 1 and intermediate dose pulsed IL-2 (SQ) on days 1-3. Patients receive low dose IL-2 (SQ) on days 4-14. Treatment may be delayed up to 7 days to allow for recovery and for tumor restaging, but daily low dose IL-2 is continued in this interval. Patients are followed at 4 weeks and then every 8 weeks until progression or death.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed nonhematologic malignancy Refractory disease or disease for which no effective standard therapy exists HER2 overexpression in tumor tissue Measurable or evaluable disease No CNS metastases Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Menopausal status: Not specified Performance status: CALGB 0-1 Life expectancy: At least 3 months Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times normal SGOT no greater than 5 times normal Alkaline phosphatase no greater than 5 times normal Renal: BUN no greater than 1.5 times normal Creatinine no greater than 1.5 times normal Cardiovascular: No uncontrolled or severe cardiac disease LVEF at least 45% by MUGA or echocardiogram Other: HIV negative No immunologic disease (e.g., autoimmune disease) Negative viral hepatitis antibodies No psychiatric conditions which would prevent compliance with treatment Not pregnant or nursing Fertile patients must use effective contraception No active uncontrolled bacterial, viral, or fungal infection Prior or concurrent malignancy allowed

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior interleukin-2 (IL-2) and/or herceptin allowed No concurrent immunosuppressive drugs or other immunomodulators (other than IL-2) Chemotherapy: At least 6 weeks since nitrosoureas, melphalan, or mitomycin More than 4 weeks since other chemotherapy Endocrine therapy: No concurrent corticosteroids Radiotherapy: More than 4 weeks since prior radiotherapy Surgery: At least 4 weeks since major surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 1997-07; Primary Completion 2000-03 (Actual); Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Toxicity | Cycle 1 1st MoAb tx (Day 7), then Day 1 of ea subsequent cycle
  toxicity of anti-Her2 MoAB given in combo w/ IL-2

SECONDARY OUTCOMES:
In vitro cytotoxicity | pre registration, days 1 & 4 ; of cycle 3, repeat prn at cycle 4
  patient PBMC and plasma with target HER2 expressing cell lines
Lymphocyte phenotyping | Days 1 & 4 of cycle 3; repeat prn in cycle 4
Anti tumor response | pre registration; post tx: q 8 wks until progression or death
  Tumor measurement

CONTACTS AND LOCATIONS:
Overall Officials: Gini Fleming, MD, Study Chair — University of Chicago
Locations (34):
- United States (34):
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vermont Cancer Center, Burlington, Vermont

REFERENCES:
- [Result] Fleming GF, Meropol NJ, Rosner GL, Hollis DR, Carson WE 3rd, Caligiuri M, Mortimer J, Tkaczuk K, Parihar R, Schilsky RL, Ratain MJ. A phase I trial of escalating doses of trastuzumab combined with daily subcutaneous interleukin 2: report of cancer and leukemia group B 9661. Clin Cancer Res. 2002 Dec;8(12):3718-27. PMID 12473581
- [Result] Fleming GF, Meropol NJ, Hollis DR, et al.: Phase I trial of recombinant human anti-Her2 monoclonal antibody (H) plus low-dose interleukin-2 (IL-2) in patients with solid tumors. [Abstract] Proceedings of the American Society of Clinical Oncology 17: A710, 1999.